CLINICAL TRIAL: NCT06137053
Title: Effect of Telitacicept on Transitional Regulatory B Cells in Patients With Systemic Lupus Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yanfeng Hou (Other)
Responsible Party: Sponsor-Investigator, Yanfeng Hou, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: ZGC2022-11-26
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Telitacicept; Systemic Lupus Erythematosus; Therapy
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: Standard treatment for SLE + Telitacicept 160 mg qw
- Control group: Standard treatment for SLE

SUMMARY:
The effect of Telitacicept treatment on the changes of transitional regulatory B lymphocyte T1, T2B cell subsets and plasma blasts and the expression levels of cytokines IL-10, IL-35, April and BAFF in SLE.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis meets the 2019 EULAR/ACR classification criteria for SLE;
2. Age 18-70 years old;
3. To be on a stable SLE regimen, participants were required to receive standard treatment at least 1 month prior to treatment with a biologic (Telitacicept);
4. Lupus activity Index score (SELENA-SLEDAI) ≥ 8 at screening;
5. Positive anti-nuclear antibody or anti-DSDNA antibody;
6. Combined antiphospholipid syndrome should meet the diagnostic criteria: that is, meet one clinical criterion and one laboratory criterion.

Exclusion Criteria:

1. Active infections (such as shingles, HIV infection, active tuberculosis, etc.) during the screening period;
2. Central nervous system disease (including epilepsy, psychosis, organic encephalopathy syndrome, cerebrovascular accident, encephalitis, central nervous system vasculitis) caused by SLE or not caused by SLE in the last 2 months;
3. Have active hepatitis or a history of severe liver disease;
4. Patients with immune deficiency, uncontrolled severe infection, and active or recurrent digestive ulcer;
5. Pregnant women, breastfeeding women and men or women who have planned to have a baby in the last 12 months;
6. Allergic reaction: history of allergic reaction to human biological products;
7. Those who received live vaccine within the last month;
8. Participants who have participated in any clinical trial within 28 days prior to initial screening/or 5 times the half-life of the study compound (taking an older time);
9. B cell targeted therapy, such as rituximab or epazumab, within one year;
10. Use tumor necrosis factor inhibitors and interleukin-receptor blockers within one year;
11. Patients receiving intravenous gamma globulin (IVIG), prednisone ≥ 100 mg/d for more than 14 days within one month or undergoing plasmapheresis;
12. Psychopaths with depression or suicidal thoughts.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with systemic lupus erythematosus meeting inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of transitional regulatory B cells | prior treatment
  "A subset of B cells, including T1 and T2 B cells, that secrete immunosuppressive factors and act as negative immune regulators.
Number of transitional regulatory B cells | After 12 weeks of treatment
  "A subset of B cells, including T1 and T2 B cells, that secrete immunosuppressive factors and act as negative immune regulators.
Number of transitional regulatory B cells | After 24 weeks of treatment
  "A subset of B cells, including T1 and T2 B cells, that secrete immunosuppressive factors and act as negative immune regulators.
Number of transitional regulatory B cells | After 36 weeks of treatment
  "A subset of B cells, including T1 and T2 B cells, that secrete immunosuppressive factors and act as negative immune regulators.

CONTACTS AND LOCATIONS:
Locations (1):
- Yanfeng Hou, Jinan, Shandong, China